CLINICAL TRIAL: NCT01035606
Title: Plasticity in Brain Network to Enhance Cognitive Rehabilitation
Brief Title: Training in Goal-directed Attention Regulation for Individuals With Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4605-I
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Brain Injury
Keywords: attention; rehabilitation; training; functional MRI; executive function; brain injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: The design for Arms 1 and 2 was a cross-over design. Half the participants completed Arm 1 first and then crossed-over to Arm 2; the remaining half completed Arm 2 first and then crossed-over to Arm 1. Thus, all participants completed both Arm 1 and 2.
  Arm 3 represented a parallel study. Participants enrolled in this arm did not cross-over to any other condition.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Goal-oriented Attention Regulation Training (Experimental): training in goal-directed attention regulation
  Interventions: Behavioral: training in goal-directed attention regulation
- Education (Active Comparator): brain health education
  Interventions: Behavioral: brain health education
- Technology-assisted Goal-directed Self-Regulation Training (Experimental): computer-assisted training in goal-directed attention regulation
  Interventions: Behavioral: computer-assisted training in goal-directed attention regulation

INTERVENTIONS:
Behavioral: training in goal-directed attention regulation — training in goal-directed attention regulation
  Arms: Goal-oriented Attention Regulation Training
Behavioral: brain health education — brain health education workshops
  Arms: Education
Behavioral: computer-assisted training in goal-directed attention regulation — computer-assisted training in goal-directed attention regulation, with trainer guidance and cognitive games to practice skills
  Arms: Technology-assisted Goal-directed Self-Regulation Training

SUMMARY:
Brain injuries affect the lives of numerous Veterans. This study examines how the brain is affected by injury and how rehabilitation training for attention dysfunction may change brain functioning.

DETAILED DESCRIPTION:
Traumatic brain injuries (TBI) are a leading cause of long-term disability among combat Veterans. The most common and persistent sequelae after TBI are cognitive-behavioral deficits in 'executive control' and 'attention' functions. Such abnormalities may directly contribute to poor long-term outcomes as well as impede rehabilitation of dysfunction in other cognitive and motor domains. Effective treatments would potentially make a major impact in improving functional outcomes, but consistently effective treatments are not available. The overall goal of this research is to improve the investigators' understanding of plasticity in brain function after TBI and to develop improved cognitive neurorehabilitation treatments. The intervention involves individual and group-based training in cognitive skills.

ELIGIBILITY:
Inclusion Criteria:

* history of traumatic brain injury
* greater than 1 week from injury
* residual dysfunction related to attention and executive control

Exclusion Criteria:

* aphasia
* active illicit drug use
* severe depression
* contraindications to MRI scanning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D'Esposito, MD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

REFERENCES:
- [Background] Novakovic-Agopian T, Chen AJ, Rome S, Abrams G, Castelli H, Rossi A, McKim R, Hills N, D'Esposito M. Rehabilitation of executive functioning with training in attention regulation applied to individually defined goals: a pilot study bridging theory, assessment, and treatment. J Head Trauma Rehabil. 2011 Sep-Oct;26(5):325-38. doi: 10.1097/HTR.0b013e3181f1ead2. PMID 21169860
- [Result] Chen AJ, Novakovic-Agopian T, Nycum TJ, Song S, Turner GR, Hills NK, Rome S, Abrams GM, D'Esposito M. Training of goal-directed attention regulation enhances control over neural processing for individuals with brain injury. Brain. 2011 May;134(Pt 5):1541-54. doi: 10.1093/brain/awr067. Epub 2011 Apr 22. PMID 21515904
- See also: Northern California Institute for Research and Education — http://www.ncire.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred for this study by their physicians and treatment providers due to history of acquired brain injury and chronic cognitive complaints involving distractibility and difficulties with problem solving, organization, and multitasking
Groups:
- Goal-oriented Attention Regulation Training: Therapist-guided training in goal-oriented attention regulation in a group format
Period: Overall Study
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training
Started | 19 | 19 | 11
Completed | 16 | 16 | 7
Not Completed | 3 | 3 | 4
Not completed — change in health, job demands,family | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training | Total
Number analyzed (Participants) | 19 | 19 | 11 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 11 | 49
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.2) | 50.4 (12.2) | 51.8 (12.0) | 51.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 0 | 20
  Male | 9 | 9 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Self-report
Description: Responses to goal processing questionnaire relating to areas of personal goal-based functioning. This scale measured participants self-perceived changes to their cognitive and emotional functioning. Participants indicated the degree to which they perceived changes to 11 questions after receiving trainings in Arm 1 and Arm 3 on a 10-point scale (1=domain became worse, 5 = no change, 10 = domain improved). Participants did not complete this measure after Arm 2.
Time Frame: 5 Weeks (After completion of active trainings in Arm 1 and Arm 3)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training
Number analyzed (Participants) | 16 | 0 | 7
units on a scale
  Stop and Relax during stressful times | 7.79 (1.39) |  | 6.49 (1.38)
  Stop and Refocus on current goals | 7.61 (1.36) |  | 7.73 (1.12)
  Divide a complex task into more manageable tasks | 7.60 (1.15) |  | 6.89 (1.26)
  Hold information in mind | 7.19 (1.06) |  | 6.83 (1.82)
  Complete tasks | 7.15 (1.44) |  | 7.3 (1.42)
  Interact in social settings | 7.08 (1.25) |  | 5.2 (0.70)
  Choose feasible daily goals to accomplish | 7.07 (1.07) |  | 6.99 (1.40)
  Prioritize | 6.96 (1.01) |  | 7.24 (1.41)
  Manage energy | 6.52 (1.16) |  | 6.29 (1.46)
  Manage distractions | 6.29 (1.23) |  | 6.47 (1.32)
  Manage anxiety | 6.16 (1.6) |  | 5.24 (1.24)

2. Secondary Outcome: Change From Baseline to Post-training for Task Errors on a Functional Performance Measure
Description: Participants completed a functional assessment task, the modified Multiple Errands Task (MET). The MET is an unstructured functional task that permits assessment of participants' abilities to follow outlined rules and complete multiple 'real-world' tasks in a limited time period. Participants were provided written instructions and a map of the hospital where the assessment took place, and were instructed to complete 12 subtasks in 40 minutes while following 9 specified rules. Participants completed this at task at baseline and following Training (Arms 1 & 2, but not 3). Outcome measure was computed as post-training - baseline (negative value reflects less errors made post-training).
Time Frame: 5 weeks (After completion of Arm 1 and Arm 2)
Measure: Mean (Standard Deviation); unit: Number of task failures
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training
Number analyzed (Participants) | 16 | 16 | 0
Number of task failures | -3.7 (2.8) | -1.8 (3.5) |
Statistical Analysis 1: Comparison: Goal-oriented Attention Regulation Training vs Education; Test type: Superiority; p < .01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change to Attention and Executive Functioning Composite Scores
Description: Participants completed the following neuropsychological measures of attention and executive functions before and after Arms 1 and 2, but not Arm 3.
  Letter Number Sequencing from WIAT-III; Auditory Consonant Trigram: 9,18, 36 seconds; Digit Vigilance Test (Time and Errors); DKEFS subtests: Design Fluency, Verbal Fluency Switching, Inhibition (Time and Errors); and Inhibition/Switching (Time and Errors); and Trails B. Performance on these measures were scored based upon age, and when available, educational and repeated administration norms. Resultant scores were transformed into z-scores and aggregated to form a composite measure. Higher z-scores reflect better functioning.
  The unit of analysis for this outcome was the change score from baseline to post-training. Positive change scores reflect improved performance over time[post-training - baseline], whereas negative change scores reflect worsening performance over time.
Time Frame: 5 weeks (After completion of Arm 1 and Arm 2)
Measure: Mean (Standard Deviation); unit: Aggregate Z-scores
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training
Number analyzed (Participants) | 16 | 8 | 0
Aggregate Z-scores | 0.82 (0.20) | 0.03 (0.11) |
Statistical Analysis 1: Comparison: Goal-oriented Attention Regulation Training vs Education; Test type: Superiority; p < .01, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Goal-oriented Attention Regulation Training | Education | Technology-assisted Goal-directed Self-Regulation Training
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/11
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/11

LIMITATIONS AND CAVEATS:
Overall, recruitment challenges resulted in small numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No